CLINICAL TRIAL: NCT06745830
Title: Lymph Node Pathologic Grading Strategy: Under the Backdrop of the IASLC Grading System for Invasive Lung Adenocarcinoma - a Retrospective Cohort Study
Brief Title: Lymph Node Pathologic Grading Strategy
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Other Study IDs: FUSCCLN1203
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Invasive LUAD who underwent surgical resection
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The percentage of high-grade patterns in metastatic LNs (mLNs) that can predict poor outcomes has yet to be determined. Additionally, the potential implications of other histologic patterns in metastatic lymph nodes on patient outcomes warrant further investigation.

We conducted a retrospective cohort study to investigate the prognostic value of pathologic pattern in metastatic lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

From January 2011 to September 2021, we consecutively collected patients with invasive LUAD who underwent surgical resection at the Department of Thoracic Surgery, Fudan University Shanghai Cancer Center.

Exclusion Criteria:

1. adenocarcinoma in situ, minimally invasive adenocarcinoma, invasive mucinous adenocarcinoma, and other variants of adenocarcinoma;
2. incomplete common driver mutation data;
3. unavailable pathologic slides.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2011 to September 2021, we consecutively collected patients with invasive LUAD who underwent surgical resection at the Department of Thoracic Surgery, Fudan University Shanghai Cancer Center.Exclusion criteria were the following: (1) adenocarcinoma in situ, minimally invasive adenocarcinoma, invasive mucinous adenocarcinoma, and other variants of adenocarcinoma; (2) incomplete common driver mutation data; and (3) unavailable pathologic slides.
Sampling Method: Non-Probability Sample
Enrollment: 2998 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
5-year RFS | 5 years

SECONDARY OUTCOMES:
5-year OS | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China